CLINICAL TRIAL: NCT00462423
Title: Abraxane and Avastin as Therapy for Patients With Malignant Melanoma, a Phase II Study
Acronym: AbraxAvast
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Lynn E. Spitler, MD (Other)
Collaborators: Celgene Corporation (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Lynn E. Spitler, MD, Director, Northern California Melanoma Center
Organization: Northern California Melanoma Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 070223
Record Dates: First submitted 2007-04-18; First posted 2007-04-19 (Estimated); Results first posted 2014-01-08 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Metastatic Malignant Melanoma
Keywords: Metastatic malignant melanoma; First-line therapy
MeSH Terms: conditions — Melanoma | interventions — Bevacizumab; Albumin-Bound Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single Arm, Open Label (Experimental): Single Arm, Open Label trial of Abraxane and Avastin
  Interventions: Drug: Avastin; Drug: Abraxane

INTERVENTIONS:
Drug: Avastin — Avastin 10 mg/kg IV every 2 weeks (without rest period).
  Other Names: Avastin: bevacizumab.
Drug: Abraxane — Abraxane 150 mg/m2 IV weekly for 3 weeks of a 28-day cycle.

SUMMARY:
The study is an open-label, single arm multicenter Phase II study to evaluate the safety and efficacy of the combination of Abraxane and Avastin as first-line therapy for patients with unresectable metastatic malignant melanoma. The patient sample will be approximately 50 individuals, males and females 18 years of age or older with measurable metastatic melanoma.

Patients will be treated with Abraxane administered weekly for 3 weeks via a 30-minute IV infusion at150 mg/m2 followed by 1 week rest (28-day cycle). Avastin will be administered in a dose of 10 mg/kg every 2 weeks (without rest period). Patients will be evaluated for disease progression every 2 months and those who do not have disease progression or unacceptable toxicity will be offered ongoing therapy until they have progressive disease or unacceptable toxicity.

DETAILED DESCRIPTION:
It has been suggested that chemotherapy administration may be synergistic with the effects of an antiangiogenic agent such as Avastin. A "Proof of Principal" of the concept of the synergistic effects of chemotherapy and antiangiogenic therapy has been shown in the favorable results reported with temozolomide administered in combination with thalidomide in melanoma, the favorable results reported for the use of FOLFOX4 in combination with Avastin in previously treated patients with advanced or metastatic colorectal cancer, and the approval of the combination of Avastin with 5-fluorouracil-based chemotherapy in the treatment of patients with metastatic carcinoma of the colon or rectum.

A number of lines of evidence suggest that the combination of Abraxane and Avastin may be effective as first-line therapy for melanoma:

* Taxanes are active agents in melanoma:

  1. In a clinical trial in patients who had failed combination chemotherapy (the Dartmouth regimen, there was a 24% response rate in patients treated with paclitaxel (in combination with tamoxifen).
  2. Paclitaxel is being used in a Phase III trial with carboplatin and Sorafenib in patients with metastatic melanoma who have failed no more than one previous systemic chemotherapeutic treatment.
  3. In a phase II trial of docetaxel in patients with metastatic melanoma, objective responses lasting more than 2 years were observed.
* Abraxane is a taxane that has efficacy superior to that of Taxol for the treatment of metastatic breast cancer. Abraxane was evaluated as first- and second-line therapy for patients with metastatic melanoma. Results were encouraging. In this study, Abraxane will be combined with Avastin in an effort to improve the clinical benefit and prolong the time to disease progression.

The primary end-point of the study is progression-free survival (PFS) at 4 months. Secondary end-points include progression-free survival, overall survival (OS), objective Response Rate (RR) in patients with measurable lesions, time to objective response, duration of objective response in patients with measurable lesions, and safety and tolerability of this combination.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed, (surgically incurable or unresectable) stage III or IV metastatic malignant melanoma..
* Must be chemo naïve. Surgical adjuvant therapy with interferon, vaccines, or cytokines is permitted. Prior adjuvant therapy with chemotherapeutic agents is not allowed. Prior therapy for metastatic disease that is not chemotherapy is allowed. Must have discontinued prior allowable therapy at least 4 weeks prior to initiation of dosing.
* A minimum of 1 measurable lesion according to RECIST criteria.
* ECOG performance status of 0-1.
* Age ≥ 18 years.
* Adequate hematologic, renal and liver function as defined by laboratory values performed within 14 days prior to initiation of dosing.
* Patients must have recovered from effects of major surgery.
* Women of childbearing potential should be using an effective method of contraception. Women of childbearing potential must have a negative urine or serum pregnancy test up to 28 days prior to commencement of dosing and be practicing medically approved contraceptive precautions for at least 6 months after completion of treatment as directed by their physician.
* Men should use an effective method of contraception during treatment and for at least 6 months after completion of treatment as directed by their physician.
* Must have recovered from all prior treatment-related toxicities to NCI CTCAE (v 3.0) Grade of 0 or 1, except for toxicities not considered a safety risk such as alopecia.
* Before study entry, written informed consent must be obtained. Written informed consent must be obtained from the patient prior to performing any study-related procedures.

Exclusion Criteria:

* Prior systemic therapy for metastatic disease with chemotherapy.
* Psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before trial entry.
* Major surgery or radiation therapy within 4 weeks of starting the study treatment.
* Known CNS disease.
* Previous Grade 2 or higher sensory neuropathy
* NCI CTCAE (V 3.0) grade 3 hemorrhage within 4 weeks of starting the study treatment.
* History of or known spinal cord compression, or carcinomatous meningitis, or evidence of symptomatic brain or leptomeningeal disease on screening CT or MRI scan.
* Any of the following within the 6 months prior to study drug administration: myocardial infarction, severe/unstable angina, coronary/peripheral artery bypass graft, symptomatic congestive heart failure, cerebrovascular accident or transient ischemic attack, or pulmonary embolism.
* Ongoing cardiac dysrhythmias of NCI CTCAE Version 3.0 grade ≥ 2.
* Inadequately controlled hypertension (defined as systolic blood pressure > 150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* Concurrent treatment on another clinical trial. Supportive care trials or non-treatment trials, e.g. QOL, are allowed.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study.
* Previous cancer (unless a DRS interval of at least 5 years) or concurrent malignancies at other sites with the exception of surgically cured carcinoma in-situ of the cervix and basal or squamous cell carcinoma of the skin.
* Known clinically uncontrolled infectious disease including HIV positivity or AIDS-related illness.
* Pregnant or nursing. Use of effective means of contraception (men and women) in subjects of child-bearing potential.
* New York Heart Association (NYHA) Grade II or greater congestive heart failure.
* Symptomatic peripheral vascular disease.
* Significant vascular disease (e.g. aortic aneurysm, aortic dissection).
* Evidence of bleeding diathesis or coagulopathy.
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0, anticipation of need for major surgical procedure during the course of the study
* Minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0
* Proteinuria at screening as demonstrated by urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥ 2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Serious, non-healing wound, ulcer, or bone fracture
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-04; Primary Completion 2011-04 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lynn E. Spitler, MD, Principal Investigator — Northern California Melanoma Center
Locations (2):
- United States (2):
  - Northern California Melanoma Center, San Francisco, California
  - The Angeles Clinic and Research Institute, Santa Monica, California

REFERENCES:
- [Background] Hurwitz H, Fehrenbacher L, Novotny W, Cartwright T, Hainsworth J, Heim W, Berlin J, Baron A, Griffing S, Holmgren E, Ferrara N, Fyfe G, Rogers B, Ross R, Kabbinavar F. Bevacizumab plus irinotecan, fluorouracil, and leucovorin for metastatic colorectal cancer. N Engl J Med. 2004 Jun 3;350(23):2335-42. doi: 10.1056/NEJMoa032691. PMID 15175435
- [Background] Gradishar WJ, Tjulandin S, Davidson N, Shaw H, Desai N, Bhar P, Hawkins M, O'Shaughnessy J. Phase III trial of nanoparticle albumin-bound paclitaxel compared with polyethylated castor oil-based paclitaxel in women with breast cancer. J Clin Oncol. 2005 Nov 1;23(31):7794-803. doi: 10.1200/JCO.2005.04.937. Epub 2005 Sep 19. PMID 16172456
- See also: Link to Northern California Melanoma Center Website — http://www.melanomacenter.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm, Open Label: Single Arm, Open Label trial of Abraxane and Avastin
  Abraxane and Avastin : Abraxane 150 mg/m2 IV weekly for 3 weeks of a 28-day cycle; Avastin 10 mg/kg IV every 2 weeks (without rest period).
Period: Overall Study
Arm/Group | Single Arm, Open Label
Started | 50
Completed | 50
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Single Arm, Open Label
Number analyzed (Participants) | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 29
  >=65 years | 21
Age, Continuous [Mean (Full Range); unit: years] | 62 (NA) [25 to 89]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 32
Region of Enrollment [Number; unit: participants]
  United States | 50

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) at 4 Months
Description: Progression-free survival at 4 months from first treatment as determined by RECIST 1.0
Time Frame: 4 months.
Measure: Number (95% Confidence Interval); unit: percentage of patients
Arm/Group | Single Arm, Open Label
Number analyzed (Participants) | 50
percentage of patients | 75 [63 to 87]

2. Secondary Outcome: Progression-free Survival
Description: Median time of progression-free survival from first treatment according to RECIST 1.0
Time Frame: From start of treatment to disease progressin; median duration of follow-up for surviving patients was 41.6 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Single Arm, Open Label
Number analyzed (Participants) | 50
Months | 7.63 [5.56 to 9.93]

3. Secondary Outcome: Overall Survival (OS)
Description: The duration of overall survival was defined as the number of months between the start date of protocol treatment and the date of death (irrespective of cause), and was right-censored at the date of last contact for patients who were alive as of the data cutoff.
Time Frame: April 2007 through December 2010
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Single Arm, Open Label
Number analyzed (Participants) | 50
months | 16.8 [12.6 to 20.7]

4. Secondary Outcome: Objective Response Rate (RR) in Patients With Measurable Lesions Time to Objective Response
Description: The objective response rate is defined as the percentage of patients showing complete or partial response.
Time Frame: The median duration of follow-up for surviving patients was 41.6 months.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Single Arm, Open Label
Number analyzed (Participants) | 50
Percentage of participants | 36 [23 to 51]

5. Secondary Outcome: Safety and Tolerability of This Combination
Description: See adverse events Table
Time Frame: April 2007 through December 2010
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 years.
Arm/Group | Single Arm, Open Label
Serious Adverse Events (participants affected / at risk) | 13/50
Other Adverse Events (participants affected / at risk) | 11/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm, Open Label (N=50)
Atrial Flutter (Cardiac disorders) | 1 (1) — Grade 3
Hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Grade 3
Small intestinal perferation (Gastrointestinal disorders) | 1 (1) — Grade 3
Supraventricular tachycardia (Cardiac disorders) | 1 (1) — Grade 3
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) — Grade 3
Transient ischemic attack (Nervous system disorders) | 1 (1) — Grade 3
Pulmonary embolism (Blood and lymphatic system disorders) | 1 (1) — Grade 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Grade 3
Renal tubular necrosis (Renal and urinary disorders) | 1 (1) — Grade 3
Bowel perforation (Gastrointestinal disorders) | 1 (1) — Grade 3
Palmar-plantar erythrodysesthesia (Musculoskeletal and connective tissue disorders) | 1 (1) — Grade 3
Macular edema (Eye disorders) | 1 (1) — Grade 3
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm, Open Label (N=50)
Peripheral neuropathy (Nervous system disorders) | 5 (5) — Grade 3 - 4
Neutropenia (Blood and lymphatic system disorders) | 6 (6) — Grade 3 - 4.

LIMITATIONS AND CAVEATS:
This was a single arm study. Follow-up trials to further explore this regimen are warranted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less